CLINICAL TRIAL: NCT06870968
Title: An Exercise Training Intervention for Depressive Symptoms in Youth With MS: A Randomized Controlled Feasibility Trial
Brief Title: FIT-ATOMIC Exercise Feasibility Trial
Acronym: FIT-ATOMIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: National Multiple Sclerosis Society (Other); Multiple Sclerosis Society of Canada (Other); University of California, San Diego (Other); Children's Hospital of Philadelphia (Other); Alberta Health Services, Calgary (Other); Queen's University (Other); University of Illinois at Chicago (Other); Unity Health Toronto (Other)
Responsible Party: Principal Investigator, E. Ann Yeh, Staff Neurologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1000080992
Record Dates: First submitted 2024-09-12; First posted 2025-03-11 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-09

CONDITIONS: Neuroinflammatory Diseases; Multiple Sclerosis
Keywords: multiple sclerosis; physical activity; depression; exercise intervention; biomarkers; irisin; brain-derived neurotrophic factor BDNF; randomized controlled trial; feasibility study; home-based exercise; youth; children; pediatric; brain and mental health
MeSH Terms: conditions — Neuroinflammatory Diseases; Multiple Sclerosis; Motor Activity; Depression; Psychological Well-Being | interventions — Exercise; Range of Motion, Articular

STUDY DESIGN:
Intervention Model Description: Participants will be randomized at the time of enrolment to either an Exercise Training group or a Mobility and Flexibility Training group.
Who Masked: Participant, Outcomes Assessor
Masking Description: To avoid bias or influence in outcomes, participants will not be informed which training group is the intervention group and which is the sham/control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Training Group (Active Comparator): The exercise training will follow a progressive interval-based training program designed for youth with MS. Participants will engage in three weekly exercise sessions. Participants will be given access to links to live virtual structured exercise sessions. The sessions will be scheduled weekly in partnership with a coach. A trained fitness instructor will lead the participants in a 10-minute warm-up, followed by 30 minutes of interval training, and a 10-minute stretching and cool down activity. Intervals will progress in intensity over the course of the 20-week program and progression will be based on individualized target heart rate zones established from baseline exercise testing.
  Interventions: Behavioral: Exercise Training
- Mobility & Flexibility Training Group (Sham Comparator): The Mobility & Flexibility Training Program focuses on mobility and flexibility. The training will be focused on improving mobility and flexibility through three times a week stretching and mobility program. A 5-minute warm up will be followed by a series of stretches and mobility patterns that will be repeated as a circuit four times. Each session will focus on a specific muscle group - upper body, lower body or core. The classes will be led by a fitness instructor in the same manner as the exercise group with a virtual link sent to the participants.
  Interventions: Behavioral: Mobility and Flexibility Training

INTERVENTIONS:
Behavioral: Exercise Training — The Exercise Training will follow a progressive interval-based training program designed for youth with MS. Participants will engage in three weekly exercise sessions. Participants will be given access to links to live virtual structured exercise sessions. The sessions will be scheduled weekly in partnership with a coach. A trained fitness instructor will lead the participants in a 10-minute warm-up, followed by 30 minutes of interval training, and a 10-minute stretching and cool down activity. Intervals will progress in intensity over the course of the 20-week program and progression will be based on individualized target heart rate zones. The session will be delivered via a live feed in order to foster social support from the participants peers enrolled in the program. Participants will have the option of completing the class in real-time and make up classes will also be available through a repository of sessions accessible through links to the repository cloud.
  Other Names: Exercise Program for Youth with MS
  Arms: Exercise Training Group
Behavioral: Mobility and Flexibility Training — The Mobility and Flexibility Training will be focused on improving mobility and flexibility through three times a week stretching and mobility program. A 5-minute warm up will be followed by a series of stretches and mobility patterns that will be repeated as a circuit four times. Each session will focus on a specific muscle group - upper body, lower body or core. The classes will be led by a fitness instructor in the same manner as the exercise intervention arm with a virtual link sent to the participants.
  Other Names: Mobility and Flexibility Training Program
  Arms: Mobility & Flexibility Training Group

SUMMARY:
This multi-center, randomized controlled feasibility trial will assess a 20-week home-based exercise intervention in youth with Multiple Sclerosis (MS). The goal is to determine the feasibility of conducting a larger, definitive trial on exercise training as a non-pharmacological approach to improve disease outcomes in this population.

Participants will be randomized to either an Exercise Training group or a Mobility and Flexibility Training group. The investigators will evaluate differences between the two groups in physical activity levels, mediators of physical activity, and psychosocial outcomes. Assessments, including clinical exams, brain MRI, eye tracking, cognitive testing, blood draws, and questionnaires, will occur at baseline and after 20 weeks. Accelerometry will be done at baseline, 10 weeks, and 20 weeks to track physical activity.

The primary objectives are to assess the feasibility of recruiting, retaining, and randomizing youth with MS and to evaluate adherence to the exercise intervention and coaching sessions. Exploratory objectives include examining changes in depressive symptoms, cognitive function, blood biomarkers (BDNF and irisin), brain volume, and fitness levels in response to the intervention.

Approximately 40 participants will be enrolled from four sites in Canada and the United States.

Primary outcomes include feasibility, acceptability, and fidelity measures. Exploratory outcomes include blood biomarkers, brain MRI, cognitive testing, and other neuropsychological measures.

DETAILED DESCRIPTION:
Overview: This research study explores the potential of exercise as a non-pharmacological treatment for youth with Multiple Sclerosis (MS). The investigators are conducting a 20-week home-based exercise program to determine if it is feasible to implement this type of intervention in a larger trial in the future. Our ultimate goal is to understand how exercise might help improve both physical and mental health outcomes for youth with MS.

Why This Study is Important: Multiple Sclerosis is a chronic disease that affects the brain and spinal cord, often leading to issues with movement, balance, vision, and other body functions. In young people, MS can have a significant impact on daily life, including mental health and cognitive abilities (such as memory and problem-solving). Medications can help manage symptoms, but there is growing interest in non-medication approaches, like exercise, to enhance the overall well-being of youth with MS. This study aims to investigate whether a structured exercise program can benefit physical fitness, mental health, and brain function in young people living with MS.

Study Design: This feasibility trial will enroll approximately 40 participants from four different locations in Canada and the United States. These participants will be youth diagnosed with MS.

Participants will be randomly assigned to one of two groups:

1. Exercise Training Group: Participants will follow a 20-week home-based exercise program, which includes structured exercises designed to improve physical fitness.
2. Mobility and Flexibility Training: Participants in this group will follow a 20-week program focused on mobility and flexibility exercises.

The study will collect data through various assessments, including:

* Clinical Exams: To monitor physical health and MS-related symptoms.
* Brain MRI: To measure changes in brain structure.
* Eye Tracking (SickKids participants only): To assess brain activity and cognitive functions.
* Cognitive Testing: To evaluate memory, attention, and other cognitive abilities.
* Blood Draws: To measure blood biomarkers related to brain health, such as Brain-Derived Neurotrophic Factor (BDNF) and irisin, which are proteins thought to be linked to exercise benefits.
* Questionnaires: To gather information on mental health, including levels of depression and overall well-being.
* Accelerometry: To measure physical activity levels throughout the study.

What the Investigators Hope to Learn: The main goal of this study is to see whether it is practical to run a large-scale trial using a home-based exercise program for youth with MS. The investigators will look at whether it is possible to successfully recruit, retain, and engage participants in the program and how well they adhere to the exercise plan.

In addition to feasibility, the study has several exploratory objectives:

1. Mental Health: The investigators want to see if participants in the exercise group show improvements in depressive symptoms compared to the control group.
2. Cognition: The investigators will evaluate whether exercise has a positive effect on thinking skills, such as memory and attention.
3. Brain Health: Through brain MRI scans, the investigators will examine whether exercise protects or enhances brain volume in areas linked to MS.
4. Fitness Levels: The investigators will measure if participants improve their physical fitness as a result of the exercise program.
5. Biomarkers: The investigators will study how exercise impacts blood levels of BDNF and irisin, which may provide insight into the biological mechanisms behind the benefits of exercise.

Why It Matters: This study is a critical first step in determining if exercise can be a viable and effective way to improve the lives of youth with MS. If successful, the findings will pave the way for a larger trial that could lead to new, non-medication-based treatments to improve mental health, cognitive function, and overall well-being in young people with MS.

By addressing the gaps in understanding how exercise benefits youth with MS, this research could offer valuable insights into developing better care strategies for this population. The results will inform not only how future exercise programs are designed but also provide a deeper understanding of the biological mechanisms linking physical activity to brain health and mood in youth with MS.

Study Locations: The study will take place across four sites:

* SickKids (Toronto, Canada)
* Stollery Children's Hospital (Edmonton, Canada)
* Children's Hospital of Philadelphia (Philadelphia, USA)
* University of California, San Diego (San Diego, USA)

How This Study Will Help in the Future: The information the investigators gather from this feasibility trial will help shape a larger, more definitive study to further explore whether exercise can be widely implemented as a safe and effective treatment option for youth with MS. It could lead to new therapeutic strategies that do not rely solely on medication but focus on holistic approaches to health and wellness.

ELIGIBILITY:
Inclusion Criteria:

* Youth and young adults 11-25 years of age
* MS diagnosis or clinically isolated syndrome per revised McDonald diagnostic criteria and International Pediatric MS Study Group Criteria
* A score of 10 or above on the CES-DC scale.

Exclusion Criteria:

* Have non-specific white matter abnormalities and metabolic or infectious etiologies for white matter abnormalities
* Do not speak and read English at a level needed to complete the questionnaires (4th grade level)
* Have significant motor disability (EDSS ≥4)
* Are at increased risk of cardiac or other complications of exercise testing, as determined by the pediatric neurologist or physician

Ages: 11 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Participant accrual rate | From enrollment to the end of study
  Number of participants enrolled per year
Fidelity of delivering the intervention | From enrollment to the end of intervention at 20 weeks
  ASPIRE fidelity coaching checklist. This measure assesses the fidelity with which study coaches deliver the intervention during calls with participants. Participants are scored on a scale from 0 to 2, based on the extent to which the intervention components are covered:
  0: Did not cover - The intervention component was not addressed during the call.
  1. Partially covered - The intervention component was addressed to some extent, but not fully.
  2. Fully covered - The intervention component was fully addressed, meeting the intended criteria for delivery.
  A higher score reflects a more complete and accurate delivery of the intervention as planned.
Participant drop-out rate | From enrollment to the end of study
  Percentage of total patients that dropped out of study.
Adverse event rate | From enrollment to the end of study
  Number of adverse events per total participants
Completion rate of study measures | From enrollment to the end of study
  Percentage of total patients that completed the study measures.

OTHER OUTCOMES:
Blood myokine irisin measurement | From enrollment to the end of intervention at 20 weeks
  Change in blood irisin levels (ng/mL) between baseline and end of 20-week intervention.
Blood brain-derived neurotrophic factor (BDNF) measurement | From enrollment to the end of intervention at 20 weeks
  Change in blood BDNF levels (ng/mL) between baseline and end of 20-week intervention.
Change in brain volumes | From enrollment to the end of intervention at 20 weeks
  This outcome measure assesses changes in brain volume following the intervention. MRI scans of the brain will be performed at baseline and at 20 weeks. The outcome metrics include the absolute change in brain volume (mm^3), percentage change in brain volume, and variance in brain volume changes across participants.
Cognitive flexibility - Dimensional Change Card Sort test | From enrollment to the end of intervention at 20 weeks
  This outcome measure evaluates cognitive performance based on a combination of accuracy and reaction time. The scoring process combines accuracy and reaction time, using a 2-vector system where each vector is scored from 0 to 5. The final score ranges from 0 to 10. If a participant's accuracy is 80% or lower, the final score is based solely on accuracy. If accuracy exceeds 80%, both accuracy and reaction time are combined to calculate the final score. A score below 4 indicates that accuracy was insufficient (lower than or equal to 80%) to allow for a reaction time score. Higher scores are associated with better cognitive flexibility. Normative data are used to compare the participant's performance to age- and education-based averages, providing a contextual understanding of individual scores.
Executive function (Inhibitory control and attention) - Flanker test | From enrollment to the end of intervention at 20 weeks
  The scoring method for the Flanker test is identical to that of the DCCS and uses a 2-vector scoring system based on accuracy and reaction time, each scored on a scale from 0 to 5. The final computed score ranges from 0 to 10, representing the participant's overall performance. If a participant's accuracy is 80% or lower, the final computed score is based solely on accuracy. If accuracy exceeds 80%, the reaction time score and accuracy score are combined to calculate the final score. A computed score below 4 indicates that the participant did not achieve sufficient accuracy (lower than or equal to 80%) to include a reaction time component. Higher scores reflect better attention and the ability to ignore distractions, indicating stronger cognitive control. Normative data are used to compare the participant's performance to age- and education-based averages, providing a contextual understanding of individual scores.
Information Processing Speed - Oral Symbol Digit Test (OSD) | From enrollment to the end of intervention at 20 weeks
  The OSD assesses information processing speed, attention, and cognitive efficiency by requiring participants to match numbers with corresponding symbols using a reference key within a 120-seconds time limit. The test is scored based on the total number of correct responses (raw score), with higher scores indicating better performance.
  Changes in raw scores between Time 1 and Time 2 reflect improvements or declines in cognitive processing speed over time. Normative data are used to compare the participant's performance to age- and education-based averages, providing context for individual scores.
Free viewing eye tracking - Saccades | From enrollment to the end of intervention at 20 weeks
  This outcome measure evaluates visual attention, cognitive processing, and arousal through key eye-tracking metrics collected during free-viewing tasks. Data are recorded and analyzed to understand participants' visual and cognitive engagement with presented stimuli. The mean saccade rate (MSR) will be calculated as the frequency of macro-saccades (saccades with an amplitude of greater than or equal to 2 degress) across all videos combined.
Free viewing eye tracking - Fixations | From enrollment to the end of intervention at 20 weeks
  This outcome measure evaluates visual attention, cognitive processing, and arousal through key eye-tracking metrics collected during free-viewing tasks. Data are recorded and analyzed to understand participants' visual and cognitive engagement with presented stimuli.The mean fixation duration (MFD) will be calculated as the average time spent fixating between any two successive saccades across all video clips.
PedsQL Core Module | From enrollment to the end of intervention at 20 weeks
  This measure evaluates the health-related quality of life (HRQoL) in children and adolescents using the Varni Pediatric Quality of Life Inventory (PedsQL) Core Module. The PedsQL consists of 23 items across four dimensions: Physical, Emotional, Social, and School Functioning. Each item is scored on a 5-point Likert scale, with responses reverse-scored and transformed to a 0-100 scale, where higher scores indicate better HRQoL.
Varni Pediatric Multidimensional Fatigue Scale (PedsQL-MFS) | From enrollment to the end of intervention at 20 weeks
  The Varni Pediatric Multidimensional Fatigue Scale (PedsQL-MFS) is a tool designed to measure fatigue in children and adolescents, assessing its impact on daily functioning. The scale includes 18 items across three domains: General Fatigue, Sleep/Rest Fatigue, Cognitive Fatigue. Participants rate their level of fatigue over the past month on a 5-point Likert scale, where higher scores indicate less fatigue. Items are reverse-scored and transformed to a 0-100 scale, with higher scores representing less fatigue. Subscale scores are calculated for each dimension, and a total fatigue score is derived by averaging the scores from all three domains.
The Centre for Epidemiological Studies Depression Scale Children's Rating Scale (CES-DC) | From enrollment to the end of intervention at 20 weeks
  The Centre for Epidemiological Studies Depression Scale Children's Rating Scale (CES-DC) is a widely used tool for assessing depressive symptoms in children and adolescents. The scale consists of 20 items that measure symptoms of depression experienced during the past week. These symptoms are related to mood, behavior, and physical well-being, and include feelings of sadness, irritability, social withdrawal, and changes in sleep or appetite. Each item is rated on a 4-point Likert scale ranging from 0 (Not At All) to 3 (A Lot). The total score is obtained by summing the ratings across all 20 items, with higher scores indicating more severe depressive symptoms.
Screen for Anxiety-Related Disorders (SCARED) | From enrollment to the end of intervention at 20 weeks
  The Screen for Anxiety-Related Disorders (SCARED) is a self-report tool designed to screen for anxiety symptoms in children and adolescents. The scale consists of 41 items that assess symptoms related to various anxiety disorders, including generalized anxiety disorder, separation anxiety disorder, social anxiety disorder, and specific phobias. Each item is rated on a 3-point Likert scale: 0 (Not true or hardly ever true), 1 (Somewhat true or sometimes true), and 2 (Very true or often true). The total score is derived by summing the ratings across all items, with higher scores indicating more severe anxiety symptoms.
Godin Leisure-Time Exercise Questionnaire (GLTEQ) | From enrollment to the end of intervention at 20 weeks
  The GLTEQ is a self-report tool used to assess the frequency and intensity of physical activity during leisure time. The GLTEQ consists of three questions that measure the frequency of strenuous, moderate, and light physical activities performed for at least 15 minutes during a typical week.
  Participants are asked to report the number of times they engage in each level of activity over the past week, using the following intensity categories: Strenuous activity, Moderate activity, and Light activity. Each question is rated on a 4-point scale: 0 (None), 1 (once a week), 2 (twice a week), and 3 (3 or more times a week). The GLTEQ provides a score by multiplying the frequency of each activity level by a corresponding factor (9 for strenuous, 5 for moderate, and 3 for light), and then summing the results. The final score represents the overall level of physical activity, with higher scores indicating greater levels of leisure-time physical activity.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - University of California, San Diego, La Jolla, California
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Canada (2):
  - Stollery Children's Hospital, Edmonton, Alberta
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Background] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374
- [Background] Krupp LB, Banwell B, Tenembaum S; International Pediatric MS Study Group. Consensus definitions proposed for pediatric multiple sclerosis and related disorders. Neurology. 2007 Apr 17;68(16 Suppl 2):S7-12. doi: 10.1212/01.wnl.0000259422.44235.a8. PMID 17438241
- [Background] Stephens S, Schneiderman JE, Finlayson M, Berenbaum T, Motl RW, Yeh EA. Feasibility of a theory-informed mobile app for changing physical activity in youth with multiple sclerosis. Mult Scler Relat Disord. 2022 Feb;58:103467. doi: 10.1016/j.msard.2021.103467. Epub 2021 Dec 20. PMID 34954651
- [Background] Motl RW, Backus D, Neal WN, Cutter G, Palmer L, McBurney R, Schmidt H, Bethoux F, Hebert J, Ng A, McCully KK, Plummer P. Rationale and design of the STEP for MS Trial: Comparative effectiveness of Supervised versus Telerehabilitation Exercise Programs for Multiple Sclerosis. Contemp Clin Trials. 2019 Jun;81:110-122. doi: 10.1016/j.cct.2019.04.013. Epub 2019 Apr 22. PMID 31022481
- [Background] Stephens S, Berenbaum T, Finlayson M, Motl RW, Yeh EA. Youth with multiple sclerosis have low levels of fitness. Mult Scler. 2021 Sep;27(10):1597-1605. doi: 10.1177/1352458520974360. Epub 2020 Nov 27. PMID 33245672
- [Background] Bilek F, Cetisli-Korkmaz N, Ercan Z, Deniz G, Demir CF. Aerobic exercise increases irisin serum levels and improves depression and fatigue in patients with relapsing remitting multiple sclerosis: A randomized controlled trial. Mult Scler Relat Disord. 2022 May;61:103742. doi: 10.1016/j.msard.2022.103742. Epub 2022 Mar 15. PMID 35349884
- [Background] Spalletta G, Piras F, Caltagirone C, Fagioli S. Hippocampal multimodal structural changes and subclinical depression in healthy individuals. J Affect Disord. 2014 Jan;152-154:105-12. doi: 10.1016/j.jad.2013.05.068. Epub 2013 Jun 22. PMID 23800444
- [Background] Nabkasorn C, Miyai N, Sootmongkol A, Junprasert S, Yamamoto H, Arita M, Miyashita K. Effects of physical exercise on depression, neuroendocrine stress hormones and physiological fitness in adolescent females with depressive symptoms. Eur J Public Health. 2006 Apr;16(2):179-84. doi: 10.1093/eurpub/cki159. Epub 2005 Aug 26. PMID 16126743
- [Background] Wrann CD, White JP, Salogiannnis J, Laznik-Bogoslavski D, Wu J, Ma D, Lin JD, Greenberg ME, Spiegelman BM. Exercise induces hippocampal BDNF through a PGC-1alpha/FNDC5 pathway. Cell Metab. 2013 Nov 5;18(5):649-59. doi: 10.1016/j.cmet.2013.09.008. Epub 2013 Oct 10. PMID 24120943
- [Background] Cotman CW, Berchtold NC, Christie LA. Exercise builds brain health: key roles of growth factor cascades and inflammation. Trends Neurosci. 2007 Sep;30(9):464-72. doi: 10.1016/j.tins.2007.06.011. Epub 2007 Aug 31. PMID 17765329
- [Background] Erickson KI, Voss MW, Prakash RS, Basak C, Szabo A, Chaddock L, Kim JS, Heo S, Alves H, White SM, Wojcicki TR, Mailey E, Vieira VJ, Martin SA, Pence BD, Woods JA, McAuley E, Kramer AF. Exercise training increases size of hippocampus and improves memory. Proc Natl Acad Sci U S A. 2011 Feb 15;108(7):3017-22. doi: 10.1073/pnas.1015950108. Epub 2011 Jan 31. PMID 21282661
- [Background] Parrish JB, Weinstock-Guttman B, Smerbeck A, Benedict RH, Yeh EA. Fatigue and depression in children with demyelinating disorders. J Child Neurol. 2013 Jun;28(6):713-8. doi: 10.1177/0883073812450750. Epub 2012 Jul 17. PMID 22805247
- [Background] Longoni G, Brown RA, Aubert-Broche B, Grover SA, Branson HM, Fetco D, Bar-Or A, Marrie RA, Motl RW, Collins DL, Narayanan S, Arnold DL, Banwell B, Yeh EA. Physical activity and dentate gyrus volume in pediatric acquired demyelinating syndromes. Neurol Neuroimmunol Neuroinflamm. 2018 Sep 6;5(6):e499. doi: 10.1212/NXI.0000000000000499. eCollection 2018 Nov. PMID 30211252
- [Background] Grover SA, Sawicki CP, Kinnett-Hopkins D, Finlayson M, Schneiderman JE, Banwell B, Till C, Motl RW, Yeh EA. Physical Activity and Its Correlates in Youth with Multiple Sclerosis. J Pediatr. 2016 Dec;179:197-203.e2. doi: 10.1016/j.jpeds.2016.08.104. Epub 2016 Oct 4. PMID 27717498
- [Background] Stephens S, Shams S, Lee J, Grover SA, Longoni G, Berenbaum T, Finlayson M, Motl RW, Yeh EA. Benefits of Physical Activity for Depression and Fatigue in Multiple Sclerosis: A Longitudinal Analysis. J Pediatr. 2019 Jun;209:226-232.e2. doi: 10.1016/j.jpeds.2019.01.040. Epub 2019 Mar 14. PMID 30878208